CLINICAL TRIAL: NCT04310618
Title: Characterization of Mucus Solids Concentration in Patients With Bronchiectasis: Cross-sectional Study
Brief Title: Mucus Solids Concentration in Patients With Bronchiectasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad San Jorge (Other)
Collaborators: Hospital Clinic of Barcelona (Other); Asociación Murciana de Fibrosis Quistica (Unknown); University of North Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: wt%_S vs IN; Antonio Dupla Abadal 2018 (Other Grant/Funding Number: Sociedad Aragonesa de Aparato Respiratorio (SADAR))
Record Dates: First submitted 2020-02-25; First posted 2020-03-17 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-01

CONDITIONS: Bronchiectasis
Keywords: Mucus concentration
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with bronchiectasis: Adult subjets diagnosed with bronchiectasis by high-resolution computed tomography with symptomatology in stable phase
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
There is a need for biomarkers that can rapidly and sensitively detect therapeutic benefits of therapies designed to "rehydrate" airways and monitor disease severity and progression. In this study the investigators will evaluate the stability of mucus concentration in patients with bronquiectasis (CF and NCBF) and its ability to respond to acute exacerbations in order to assess whether it can be a good candidate for biomarker.

DETAILED DESCRIPTION:
Prospective cross-sectional study of repeated measurements. The recruitment will be performed in 3 different cities of Spain: Zaragoza, Barcelona and Murcia.

Subjects will be asked to repeatedly collect spontaneous and induced sputum samples in both stable and exacerbated conditions. All samples will be collected autonomously by patients in their homes after they have been instructed and supervised. Hypertonic saline nebulization will be used for sputum induction.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF (confirmed genetics) or diagnosis of non-CF bronchiectasis through high resolution computed tomography.
* Aged ≥ 18 years.
* Clinically stable at the time of recruitment.
* Chronic sputum production (able to produce spontaneous sputum daily).
* Current hypertonic saline user.
* Able to provide written informed consent and perform the trial.

Exclusion Criteria:

* Current smoker or >10 pack-year history of tobacco use.
* Patient in transplantation or retransplantation list.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with bronchiectasis
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2020-12-21 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Inter-sample variability of sputum concentration (% solids) | 2 stable weeks
  % solids will be calculated by measuring the wet to dry sputum weight ratio

SECONDARY OUTCOMES:
Inter-sample variability of sputum concentration (% solids) | 1 stable day (at 9:00 am, 12:00 am and 17:00 pm)
  % solids will be calculated by measuring the wet to dry sputum weight ratio
Sputum concentration (% solids) during the first exacerbation after recruitment | 1 day
  % solids will be calculated by measuring the wet to dry sputum weight ratio
Sputum concentration (% solids) one month after the first exacerbation after recruitment | 1 day
  % solids will be calculated by measuring the wet to dry sputum weight ratio
Forced expiratory volume at 1 second | Baseline
  Simple spirometry
Forced vital capacity | Baseline
  Simple spirometry:
Forced expiratory flow 25-75 | Baseline
  Simple spirometry
Quality of life related to cough | Baseline
  Leicester Cough Questionnaire (LCQ). Self-administered questionnaire that evaluates the impact of cough in three domains: physical, psychological, and social (each one ranged 1 to 7). It is composed of 19 questions and the "total score (range 3 to 21) is calculated by adding the domain scores together". The lower the score, the greater the severity.
Impact of cough and sputum symptoms of everyday life | Baseline
  Cough and Sputum Assessment Questionnaire (CASA-Q). Self-administered questionnaire that consists of 20 questions organized in four domains (cough symptoms, cough impact, sputum symptoms, and sputum impact). Each domain is ranged from 0 to 100. The total score is expressed over 100 and calculated doing an average of the four domains. The lower the score, the greater the severity.
Breathlessness | Baseline
  Modified Medical Research Council breathlessness scale: self-rating tool to measure the degree of disability that breathlessness poses on day-to-day activities on a scale from 0 to 4: 0, no breathlessness except on strenuous exercise; 1, shortness of breath when hurrying on the level or walking up a slight hill; 2, walks slower than people of same age on the level because of breathlessness or has to stop to catch breath when walking at their own pace on the level; 3, stops for breath after walking ∼100 m or after few minutes on the level; and 4, too breathless to leave the house, or breathless when dressing or undressing.
Ease of coughing up | Baseline
  Visual analog scales are 10-cm lines anchored at the ends by words that define the bounds of ease of coughing up options; corresponding 0 to "expectorate is very easy" and 10 to "expectorate is very difficult".
Ease of coughing up | During the first exacerbation after recruitment
  Visual analog scales are 10-cm lines anchored at the ends by words that define the bounds of ease of coughing up options; corresponding 0 to "expectorate is very easy" and 10 to "expectorate is very difficult".
Sputum colour | Baseline
  Sputum colour chart (Murray MP et al.)
Sputum colour | During the first exacerbation after recruitment
  Sputum colour chart (Murray MP et al.)
Exacerbation frequency | 12 months before enrollement
  Number of exacerbations

CONTACTS AND LOCATIONS:
Overall Officials: Marta San Miguel Pagola, Principal Investigator — Universidad San Jorge
Locations (1):
- Marta San Miguel Pagola, Zaragoza, Aragon, Spain

REFERENCES:
- See also: Sputum colour chart (Murray MP et al.) — https://www.ncbi.nlm.nih.gov/pubmed/19648517